CLINICAL TRIAL: NCT06662643
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial Comparing Staged Turnbull-Cutait Pull-through Anastomosis With Direct Anastomosis Plus Prophylactic Ileostomy in the Treatment of Low Rectal Cancer After Internal Sphincter Resection
Brief Title: A Clinical Trial Comparing Staged Turnbull-Cutait Pull-through Anastomosis With Direct Anastomosis Plus Prophylactic Ileostomy in the Treatment of Low Rectal Cancer After Internal Sphincter Resection
Acronym: STAR-TAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Collaborators: Ezhou Central Hospital (Unknown); Jingzhou Central Hospital (Other); Taihe Hospital (Other); Hubei University of Medicine (Other); Qilu Hospital of Shandong University (Other); Beijing Chao Yang Hospital (Other); Tianmen First People's Hospital (Unknown); Xiangyang Central Hospital (Other); First People's Hospital of Xianyang (Other); Central Hospital of Xiaogan (Other); Yichang Central People's Hospital (Other); Yichang Second People's Hospital (Other); Rocket Force Special Medical Center of the People's Liberation Army (Unknown); Huashan Hospital (Other)
Responsible Party: Principal Investigator, Congqing Jiang, Head of department of colorectal and anal surgery, Zhongnan Hospital of Wuhan University, Zhongnan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zhongnan Hospital Wuhan; 2024054 (Other: Zhongnan Hospital Institutional Review Board (IRB))
Record Dates: First submitted 2024-10-22; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Rectal Cancer; Rectal Carcinoma
Keywords: Low Rectal Cancer; Turnbull-Cutait; Pull-through; Internal Sphincter Resection
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staged Turnbull-Cutait Pull-through anastomosis group (Experimental): Participants in this group will undergo staged Turnbull-Cutait pull-through anastomosis for the treatment of low rectal cancer after internal sphincter resection.
  Interventions: Procedure: Delayed transanal pull-through anastomosis
- Direct anastomosis plus protective ileostomy group (Active Comparator): Participants in this group will receive direct anastomosis combined with a prophylactic ileostomy.
  Interventions: Procedure: Direct Anastomosis Plus Prophylactic Ileostomy

INTERVENTIONS:
Procedure: Delayed transanal pull-through anastomosis — Laparoscopic surgery is recommended. A standard 5-port method is used to create pneumoperitoneum after placing the trocar. The sigmoid colon and upper rectal mesentery are dissected along Toldt's fascia. Autonomic nerves should be preserved, and high ligation of the inferior mesenteric vessels with lymph node dissection is recommended. TME: Using a posterior-to-anterior approach, the mesorectal plane is dissected down to the pelvic floor, cutting the Waldeyer's fascia to enter the intersphincteric space, where sharp dissection is carried out toward the levator ani muscle hiatus. The dissection endpoint is the dentate line, where the proximal colon is exteriorized by at least 2 cm and sutured to the anal canal with 6-8 stitches, without a protective ileostomy.Two to four weeks after the first surgery, after the colon has adhered well to the surrounding tissue, the exteriorized colon is excised (under epidural or spinal anesthesia, trimming the exteriorized colon to form the anus).
  Arms: Staged Turnbull-Cutait Pull-through anastomosis group
Procedure: Direct Anastomosis Plus Prophylactic Ileostomy — ISR is categorized into partial ISR (PISR), subtotal ISR, and total ISR (TISR). Correspondingly, the anastomosis site after coloanal anastomosis is located below the levator ani hiatus (PISR, near the dentate line; subtotal-ISR and TISR, below the dentate line).The dissection steps are the same as in the first stage of the Staged Turnbull-Cutait Pull-through Anastomosis group (TME and intersphincteric space dissection).The bowel is transected at least 1 cm below the tumor, leaving a larger segment of healthy tissue on the non-tumor side while ensuring that no more than 1/3 of the dentate line is resected to avoid impairing fecal control.Anastomosis is performed using absorbable sutures under direct visualization. A protective ileostomy is created 25-30 cm from the ileocecal valve.3 to 6 months after surgery, the ileostomy is reversed. Prior to closure, digital rectal examination, defecography, MRI, colonoscopy, and other evaluation must perform.
  Arms: Direct anastomosis plus protective ileostomy group

SUMMARY:
This study targets patients undergoing ultra-low rectal cancer surgery, which requires internal sphincter resection for sphincter-saving procedures. The study compares the staged Turnbull-Cutait Pull-through anastomosis (a delayed transanal pull-through anastomosis without a protective stoma) as the experimental group with traditional anastomosis (hand-sewn/stapled) plus protective ileostomy as the control group. The aim is to assess whether the Turnbull-Cutait Pull-through colon-anal anastomosis is non-inferior to traditional ISR surgery in terms of complications (short-term such as anastomotic leakage/dehiscence, pelvic infection, anastomotic bleeding, ischemic bowel necrosis, bowel obstruction, and long-term complications such as anastomotic stricture, perianastomotic fistula, bowel obstruction, stoma-related complications, and others), postoperative anal function, quality of life, long-term oncologic outcomes, hospital stay duration, and total hospitalization costs.

DETAILED DESCRIPTION:
In recent years, with the increasing understanding of the anatomy and physiological functions of the lower rectum, the biological behavior of rectal cancer tumors, advancements in new surgical technologies, and the application of comprehensive treatment methods, there has been growing emphasis on radical surgical procedures for low rectal cancer that balance oncological safety with anal function preservation. After undergoing total mesorectal excision for low rectal cancer and subsequent coloanal anastomosis, patients often face a high risk of anastomotic leakage and pelvic infection. Therefore, a protective ileostomy is usually performed to divert feces, providing a relatively low-perfusion environment conducive to healing for ultra-low coloanal anastomoses. In the event of an anastomotic leak, the protective stoma can mitigate infection and reduce the likelihood of secondary surgeries. Nevertheless, complications following protective ileostomy, such as dehydration, chronic renal failure, and parastomal hernia, occur at rates as high as 43% . Additionally, complications related to stoma reversal exceed 20% , all of which significantly impact patients' quality of life. Approximately one-fifth of patients with preventive stomas are unable to have their stomas reversed as planned, or may require lifelong stoma formation.

In 1961, Turnbull and Cutait independently reported surgical techniques involving transanal pull-through rectal resection and delayed manual coloanal anastomosis. From a certain perspective, this procedure is the safest reconstructive method, effectively reducing anastomotic leakage-related complications and avoiding the need for a protective stoma. In recent years, its clinical application in challenging rectal cases involving radiation proctitis, complex recto-vaginal/urethral fistulas, salvage surgeries for anastomotic leaks, and low-stage progressive rectal cancer has gained increasing attention and acceptance.In 2020, a multicenter randomized controlled study published in JAMA Surgery found that the delayed anastomosis group (avoiding protective stoma) did not increase the incidence of anastomotic leaks or other complications compared to the standard coloanal anastomosis plus ileostomy group, and exhibited comparable oncological and functional outcomes . Furthermore, a recent systematic review in 2022 included one randomized controlled trial and nine observational studies with a total of 1,743 patients. This study found that staged Turnbull-Cutait anastomosis was associated with a reduced rate of anastomotic leaks.

However, the aforementioned studies and systematic reviews on staged Turnbull-Cutait anastomosis were all based on total mesorectal excision (TME), and there is a paucity of data on postoperative anal function and quality of life following this procedure, necessitating further research. As an extreme sphincter-saving surgery, ISR is currently limited in widespread adoption due to the high incidence of postoperative complications and suboptimal functional outcomes associated with anastomoses located very close to the anal verge. To date, there is a lack of systematic studies applying the Turnbull-Cutait Pull-through anastomosis to ISR procedures. Therefore, it is highly worthwhile to conduct a multicenter prospective randomized controlled study to determine whether the modified Bacon procedure (transanal pull-through, delayed anastomosis) can serve as an effective alternative to ISR-coloanal anastomosis, achieving comparable or lower rates of postoperative complications, as well as equivalent oncological radicality and defecatory function. Such research is urgently needed in this largely unexplored field. If successfully conducted and achieving its objectives, this clinical study could provide highly valuable guidance for clinical practice. Existing reports on the application of the modified Bacon procedure in low rectal cancer are generally small-sample, single-center, retrospective studies with low levels of evidence. This study aims to provide higher-level evidence through a larger-sample, prospective, multicenter, randomized controlled design.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed high- or moderate-grade adenocarcinoma or villous adenoma with malignancy on preoperative colonoscopy; tumor located ≤ 5 cm from the anal verge; primary tumor size < 5 cm in diameter.
2. All enrolled patients require intersphincteric dissection. PISR surgery must be completed with hand-sewn (preferably) or stapled coloanal anastomosis. The anastomosis should be located near the dentate line (intraoperative photos or videos must be preserved).
3. Both male and female patients aged 18-75.
4. Non-recurrent rectal cancer.
5. No concurrent multiple primary colorectal cancers.
6. Initial staging or post-neoadjuvant therapy stage: T3 above the levator ani, T1-2 below.
7. Liver or lung oligometastases deemed resectable after evaluation by a multidisciplinary team (MDT).
8. Patients may or may not have received neoadjuvant chemoradiotherapy.
9. Patients and families must understand and be willing to participate in this study, providing written informed consent.
10. Good anal function (Wexner incontinence score ≤ 5).

Exclusion Criteria:

1. History of malignant colorectal tumors.
2. Previous colorectal or anorectal surgeries or diseases.
3. Patients requiring emergency surgery due to intestinal obstruction, perforation, or bleeding.
4. Tumor invasion into the external sphincter, levator ani, or adjacent organs requiring combined organ resection.
5. Poor preoperative anal function or incontinence (Wexner incontinence score ≥ 6).
6. History of inflammatory bowel disease (IBD) or familial adenomatous polyposis (FAP).
7. Recent diagnosis of other malignancies.
8. Participation in other clinical trials within the 4 weeks prior to enrollment.
9. ASA classification ≥ IV or ECOG performance status ≥ 2.
10. Severe hepatic, renal, cardiopulmonary, or coagulation dysfunction or serious underlying disease precluding surgery.
11. History of severe mental illness.
12. Pregnant or breastfeeding women.
13. Uncontrolled preoperative infection.
14. Other clinical or laboratory findings making the patient unsuitable for the study, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
30-Day Overall Composite Postoperative Complication Rate | postoperative 30 days
  30-day overall composite postoperative complication rate includes anastomotic leakage/dehiscence, bleeding, ischemic bowel necrosis, pelvic infection (abscess), pelvic bleeding, bowel obstruction, stoma-related complications, and other complications occurring within 30 days. Anastomotic leakage is defined according to the criteria proposed by the International Study Group of Rectal Cancer (ISREC) in 2010, graded as A, B, or C, depending on severity and management.

SECONDARY OUTCOMES:
Long-term Complications Rate | postoperative 2 years
  These include anastomotic stricture, anastomotic fistulas (e.g., rectovaginal or rectourethral fistula), bowel obstruction, stoma-related complications, inability to reverse stoma, chronic presacral sinus, and rectal prolapse (both mucosal and full-thickness).
Total Surgery Time | postoperative 1 years
  Defined as the combined time of the two stages (Phase 1 + Phase 2) of Staged Turnbull-Cutait Pull-through Anastomosis with Direct Anastomosis or intersphincteric resection (ISR) plus stoma reversal time. This also includes total hospital stay (Phase 1 + Phase 2) and total hospitalization costs (Phase 1 + Phase 2).
LARS Score Questionnaire | Every 6 months in the postoperative 3 years
  Low Anterior Resection Syndrome (LARS) Score is a tool used to assess bowel function after surgical treatment for rectal cancer, particularly following low anterior resection (LAR) procedures. The LARS score evaluates the presence and severity of bowel dysfunction, which can significantly impact the quality of life for patients.
  Minimum Value: 0 Maximum Value: 42 Interpretation: Higher scores indicate worse bowel function and greater symptoms of LARS.
Wexner Incontinence Score | Every 6 months in the postoperative 3 years
  The Wexner Incontinence Score, is a validated tool used to assess the severity of fecal incontinence in patients. The Wexner score is calculated by summing the scores from each of the categories:0: No incontinence；1-5: Mild incontinence；6-10: Moderate incontinence；11-20: Severe incontinence Minimum Value: 0 Maximum Value: 20 Interpretation: Higher scores indicate worse fecal incontinence and greater impact on quality of life.
International Prostate Symptom Score (IPSS) Questionnaire | Every 6 months in the postoperative 3 years
  The International Prostate Symptom Score (IPSS) is a widely used tool for evaluating the severity of urinary symptoms in men and helps to assess the impact of these symptoms on patients' quality of life.
  Minimum Value: 0 Maximum Value: 35 Interpretation: Higher scores indicate worse urinary symptoms and a greater impact on quality of life.
The Fecal Incontinence Quality of Life Scale (FIQL). | Every 6 months in the postoperative 3 years
  Quality of Life
International Index of Erectile Function (IIEF-5) Questionnaire | Every 6 months in the postoperative 3 years
  The International Index of Erectile Function (IIEF-5) is a widely used questionnaire designed to assess erectile function in men. IIEF-5 consists of five questions that evaluate different aspects of erectile function. Each question is scored on a scale from 0 to 5, with higher scores indicating better erectile function.
  Minimum Value: 0 Maximum Value: 25 Interpretation: Higher scores indicate better erectile function and greater sexual satisfaction.
Female Sexual Function Index (FSFI) Questionnaire | Every 6 months in the postoperative 3 years
  The Female Sexual Function Index (FSFI) is a widely used questionnaire designed to assess various dimensions of female sexual function. It is a reliable tool for identifying sexual dysfunction in women.
  Minimum Value: 2 Maximum Value: 36 Interpretation: Higher scores indicate better sexual function. A total score below 26.55 suggests the presence of sexual dysfunction.
EORTC QLQ-CR29 Questionnaire | Every 6 months in the postoperative 3 years
  The EORTC QLQ-CR29 is a specific quality of life questionnaire developed by the European Organisation for Research and Treatment of Cancer (EORTC) to assess the health-related quality of life in patients with colorectal cancer. This questionnaire is an extension of the EORTC Quality of Life Questionnaire (QLQ-C30) and is designed to evaluate the specific concerns and symptoms experienced by colorectal cancer patients.
  Number of Items: 29 Scoring Range: 0 to 100 Interpretation: Higher scores indicate better functioning for functional scales and worse symptoms for symptom scales.
3-year Disease-Free Survival (3-year DFS) | postoperative 3 years
  3-year DFS refers to the duration during which patients remain free of disease following treatment (such as surgery, chemotherapy, or radiation) for a period of three years.Expressed as a percentage, with a higher percentage indicating that a greater proportion of patients remain disease-free at the 3-year mark, suggesting that the treatment may be effective in preventing recurrence or progression.Local recurrence is defined as evidence of recurrence within the pelvic area detected through digital rectal examination, colonoscopy, CT/MRI, PET-CT, or biopsy (when necessary) and confirmed to match the histopathology of the primary tumor. Distant metastasis is defined as evidence of metastasis found outside the pelvic area, including the liver, lungs, bones, or para-aortic lymph nodes.
3-year Overall Survival (3-year OS) | postoperative 3 years
  Refers to the proportion of patients who remain alive three years after the beginning of the study period.Reported as a percentage, with a higher percentage indicating a greater proportion of patients alive at the 3-year mark, which may reflect improved survival due to the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Congqing Jiang, MD, PhD, Principal Investigator — Department of colorectal and anal surgery, Zhongnan Hospital of Wuhan University
Locations (1):
- Department of colorectal and anal surgery, Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
http://www.medresman.org.cn/login.aspx http://www.medresman.org.cn/html/resman.pdf The Clinical Research Public Management Platform (Research Manager, ResMan) is an Electronic Data Capture (EDC) system that manages the clinical trial processes and records all relevant information, including baseline data of subjects such as demographic information, baseline data collected during enrollment, implementation details during the trial, and outcome data, encapsulated in the Case Record Form (CRF). All this information is recorded online via the internet and transmitted to a central database for management. Only researchers from the study group are allowed to access and operate the trial, while project managers, sponsors, or investors of funded projects have the right to view real-time data but cannot make any changes. Researchers decide whether to disclose research result data. Once data is entered and saved, any subsequent changes are automatically displayed and tracked.
Supporting Information: Study Protocol
Time Frame: Start Date: 6 months after primary results are published End Date: Data will remain available on the platform indefinitely, with no specified end date
Access Criteria: Data will be made available to researchers who meet the following criteria: 1) possess a research plan approved by an Institutional Review Board (IRB); 2) have a clear scientific objective related to this clinical study. Researchers requesting access must submit an application, and upon approval, will receive controlled access. Data will be provided in anonymized form on a secure online data platform.
URL: http://www.medresman.org.cn/login.aspx

REFERENCES:
- [Background] La Raja C, Foppa C, Maroli A, Kontovounisios C, Ben David N, Carvello M, Spinelli A. Surgical outcomes of Turnbull-Cutait delayed coloanal anastomosis with pull-through versus immediate coloanal anastomosis with diverting stoma after total mesorectal excision for low rectal cancer: a systematic review and meta-analysis. Tech Coloproctol. 2022 Aug;26(8):603-613. doi: 10.1007/s10151-022-02601-4. Epub 2022 Mar 28. PMID 35344150
- [Background] Biondo S, Trenti L, Espin E, Bianco F, Barrios O, Falato A, De Franciscis S, Solis A, Kreisler E; TURNBULL-BCN Study Group. Two-Stage Turnbull-Cutait Pull-Through Coloanal Anastomosis for Low Rectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2020 Aug 1;155(8):e201625. doi: 10.1001/jamasurg.2020.1625. Epub 2020 Aug 19. PMID 32492131
- [Background] Portale G, Popesc GO, Parotto M, Cavallin F. Delayed Colo-anal Anastomosis for Rectal Cancer: Pelvic Morbidity, Functional Results and Oncological Outcomes: A Systematic Review. World J Surg. 2019 May;43(5):1360-1369. doi: 10.1007/s00268-019-04918-y. PMID 30690655
- [Background] Remzi FH, El Gazzaz G, Kiran RP, Kirat HT, Fazio VW. Outcomes following Turnbull-Cutait abdominoperineal pull-through compared with coloanal anastomosis. Br J Surg. 2009 Apr;96(4):424-9. doi: 10.1002/bjs.6458. PMID 19283735
- [Background] Patsouras D, Yassin NA, Phillips RK. Clinical outcomes of colo-anal pull-through procedure for complex rectal conditions. Colorectal Dis. 2014 Apr;16(4):253-8. doi: 10.1111/codi.12532. PMID 24344638
- [Background] TURNBULL RB Jr, CUTHBERTSON A. Abdominorectal pull-through resection for cancer and for Hirschsprung's disease. Delayed posterior colorectal anastomosis. Cleve Clin Q. 1961 Apr;28:109-15. doi: 10.3949/ccjm.28.2.109. No abstract available. PMID 13778709
- [Background] CUTAIT DE, FIGLIOLINI FJ. A new method of colorectal anastomosis in abdominoperineal resection. Dis Colon Rectum. 1961 Sep-Oct;4:335-42. doi: 10.1007/BF02627230. No abstract available. PMID 13882795
- [Background] Man VC, Choi HK, Law WL, Foo DC. Morbidities after closure of ileostomy: analysis of risk factors. Int J Colorectal Dis. 2016 Jan;31(1):51-7. doi: 10.1007/s00384-015-2327-2. Epub 2015 Aug 6. PMID 26245947
- [Background] Murken DR, Bleier JIS. Ostomy-Related Complications. Clin Colon Rectal Surg. 2019 May;32(3):176-182. doi: 10.1055/s-0038-1676995. Epub 2019 Apr 2. PMID 31061647
- [Background] Martin ST, Heneghan HM, Winter DC. Systematic review of outcomes after intersphincteric resection for low rectal cancer. Br J Surg. 2012 May;99(5):603-12. doi: 10.1002/bjs.8677. Epub 2012 Jan 13. PMID 22246846
- [Background] Schiessel R, Karner-Hanusch J, Herbst F, Teleky B, Wunderlich M. Intersphincteric resection for low rectal tumours. Br J Surg. 1994 Sep;81(9):1376-8. doi: 10.1002/bjs.1800810944. PMID 7953423
- [Derived] Chen W, Ding J, Xiang J, Wang Y, Han J, Ye H, Wang D, Lin B, Lei J, Wu X, Di M, Fu Y, Yang G, Qin C, Chen A, Xu J, Liu W, Jiang C; STAR-TAR study group. Staged Turnbull-Cutait pull-through anastomosis comparing with direct anastomosis plus prophylactic ileostomy in the treatment of low rectal cancer after internal sphincter resection (STAR-TAR): study protocol for a randomized controlled trial. Trials. 2025 May 22;26(1):168. doi: 10.1186/s13063-025-08845-3. PMID 40405283